CLINICAL TRIAL: NCT00853944
Title: A Randomized Controlled Trial to Determine if Sitagliptin Will Enhance Islet Graft Function When Given for 1 Year Following Transplantation
Brief Title: Effect of Sitagliptin on Graft Function Following Islet Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor withdrew funding du to lack of enrollment. Lack of enrollment was due to decrease in number of islet transplant procedures
Sponsor: University of British Columbia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, David Thompson, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H08-01947
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Islet Transplantation
Keywords: islet transplantation; type 1 diabetes; incretin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P (No Intervention): subjects take 1 tablet of placebo daily
- S (Experimental): subjects take 1 tablet of sitagliptin 100 mg daily
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: sitagliptin — Subjects receive sitagliptin 100 mg po daily from the day of islet transplant until completion of the study
  Other Names: Januvia; DPP-IV inhibitor; GLP-1
  Arms: S

SUMMARY:
Islet transplantation requires a large number of islets required to achieve insulin independence and the function of the transplanted islets progressively declines over time. Evidence from animal studies and human islets in culture suggests that increasing GLP-1 levels could help with both of these problems. This study is designed to test this hypothesis using sitagliptin in a randomized clinical trial.

DETAILED DESCRIPTION:
Hypothesis: Sitagliptin taken for 12 months after an islet infusion will significantly improve islet function compared with a control group.

Purpose: To determine if sitagliptin given at the time of an islet cell transplant (ICT) results in improved islet graft function at 3 and 12 months post-transplant.

Study design: prospective, randomized, double-blind, single-centre, placebo-controlled trial.

Sample size calculation for primary outcome.

The primary outcome (stimulated insulin secretion) is a continuous variable that is normally distributed. Our previous clamp studies show an expected standard deviation of around 20% and we wish to be able to detect an increase of 33%. The result will be calculated both with and without adjustment for the number of IE / kg that a patient has received, since the literature is not clear on this issue. Analysis will be done using a two-sided t test. Sample size is estimated using an approximation of Lehr's formula for 80% power and 2-sided significance level of 5%.

m = 16 where d = δ δ = 33%, σ = 20% d 2 σ The calculation indicates a need for 6 patients per arm or a total of 12 patients for the 2 arms.

Ability of our site to perform the study

Since starting in 2003, we have performed 75 islet infusions in 31 patients, averaging one infusion per month. We are 1 of the 4 most active sites in North America (Edmonton, Miami, Minnesota are the others). We have a list of patients activated and waiting for a suitable islet donor. We anticipate that the great majority of patients will choose to participate in this trial. We should easily be able to perform the required 12 islet infusions within 2 years. The advantage of performing this study in a single therapy is the ability to keep constant variables such as eligibility criteria for recipients and choice of immunosuppressive drugs that differ considerably between centres. This approach increases the chances that the question posed will be answered by the study.

Eligible patients Eligible patients will be those in our transplant program who are about to undergo an infusion of donor islets. Criteria for entry into our program are as described (Warnock et al Arch Surg 2005;140:735). All eligible patients will be offered a chance to enter the study. Patients will need to sign an informed consent that has been approved by the Clinical Research Ethics Board of the University of British Columbia.

Randomization and Blinding Random numbers will be computer generated and placed in opaque sealed, numbered envelopes. The ratio of sitagliptin and placebo will be 1:1. The pharmacist associated with the islet transplant team will be the only team member with knowledge of the code for sitagliptin and placebo. Randomization will be done in blocks of four. The advantage of block randomization is to allow similar distribution among groups of any changes in performance of islet transplantation, such as new immunosuppression regimens, that could arise during the course of the study. There will not be any stratification. Randomization will be done just prior to islet infusion so that patients receiving either placebo or sitagliptin will be given their medication before receiving islets.

The subject and the investigators obtaining consent, performing the transplant, providing post-transplant care and performing the hyperglycemic clamp will be blind as to whether a subject is receiving sitagliptin or placebo. The placebo will be supplied by Merck and will be identical in appearance to sitagliptin. Sitagliptin and the placebo will be stored in the VGH pharmacy.

When a subject consents to participate in the study, the investigator obtaining the consent will contact the pharmacy. The pharmacy will open the next randomization envelope and dispense the medication (sitagliptin or placebo). Ongoing supply of the medication will be provided by the pharmacy in the transplant clinic during routine follow-up visits for post-transplant care.

Patient Care

All aspects of the transplantation procedure, immunosuppressive therapy and ancillary care will be performed as described (Warnock et al Arch Surg 2005;140:735) and will be similar for all patients for the duration of the study. The indications for stopping or restarting insulin are those recommended by the metabolic monitoring committee of the Collaborative Islet Transplant Registry. This will eliminate subjective investigator judgments that could affect one of the secondary endpoints (insulin dose).

Assessment of endpoints

Primary: Maximum insulin secretory capacity will be determined by a hyperglycemic glucose clamp, performed as described (Al Ghofaili et al Transplantation 2007;83:24). This will be performed at 3 and 12 months ± 2 weeks after islet infusion, with the subject having received either sitagliptin or placebo during this period. The medication will be stopped for 48 hours before the clamp to allow washout. A positive result would suggest that sitagliptin had increased functional islet mass, not that it was acting as a short-term secretagogue. The values will be expressed both as absolute numbers and as divided by the number of IE / kg received as it is not clear from the literature which is the better measurement. A baseline fasting C peptide will be drawn prior to the islet infusion.

Secondary: Patients are followed closely post transplant to maintain tight glucose control. Insulin adjustment and glucose targets are as described. The average daily insulin requirement in the week before transplant and in the week prior to stopping the study will be used for calculation. A positive result would be consistent with either an increase in functional islet mass or stimulation or insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for > 5 years with negative C peptide, GFR > 70 ml/min, BMI ≤ 28 and non-smoker for ≥ 1 year

Exclusion Criteria:

* Known hypersensitivity to sitagliptin

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-01 (Actual)

PRIMARY OUTCOMES:
Islet function as measured by hyperglycemic clamp | 3 and 12 months ± 2 weeks after islet infusion

SECONDARY OUTCOMES:
Change in insulin requirement (absolute and % decrease from pre-transplant dose) | 1 week prior to stopping the study

CONTACTS AND LOCATIONS:
Overall Officials: David M. Thompson, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada